CLINICAL TRIAL: NCT01925144
Title: Evaluation of the Impact of Increased Gastric pH Following Omeprazole Administration on the Absorption of Baricitinib in Healthy Subjects
Brief Title: A Study of Baricitinib and Omeprazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14603; I4V-MC-JAGF (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib (Experimental): Baricitinib - 10 milligram (mg) tablet administered orally, once, on Day 1.
  Interventions: Drug: Baricitinib
- Baricitinib + Omeprazole (Experimental): Baricitinib - 10 mg tablet administered orally, once, on Day 10. Omeprazole - 40 mg capsule administered orally once daily (QD) for 8 days (Days 3 through 10).
  Interventions: Drug: Baricitinib; Drug: Omeprazole

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
Drug: Omeprazole — Administered orally
  Arms: Baricitinib + Omeprazole

SUMMARY:
The main purpose of this study is to find out how the body will react to a study drug called baricitinib when taken with another drug called omeprazole.

For each participant, this study will include 2 periods in fixed order. The study will last approximately 25 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical history and physical examination
* Women not of childbearing potential due to surgical sterilization (at least 3 months after surgical hysterectomy, bilateral oophorectomy with or without hysterectomy, or bilateral tubal occlusion/ligation) confirmed by medical history, or menopause
* Have a body mass index of 18 to 29 kilograms per square meter (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Have known allergies to baricitinib, omeprazole, related compounds, or any components of the baricitinib or omeprazole formulations, or history of significant atopy
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological (including clotting disorders), or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have an absolute neutrophil count (ANC) less than 2 × 10^9 cells per liter (L) [2000 cells/microliter (μL)] at screening or Day -1. For abnormal values, a single repeat will be allowed
* Intend to use over-the-counter or prescription medication (including drugs and substances known to alter gastric potential hydrogen (pH), such as proton pump inhibitors or over-the-counter antacid remedies and/or herbal supplements within 14 days prior to dosing and during the study (with the exception of hormone replacement therapy (HRT) and occasional paracetamol, which will be permitted at the discretion of the investigator), or intended use of vitamin supplements from Day 1 until discharge from the clinical research unit (CRU)
* Have used or intend to use any drugs or substances that are known to be substrates, inhibitors, or inducers of cytochrome P450 3A4 (CYP3A4) within 30 days prior to dosing and throughout the study
* Are unable to tolerate or unwilling to undergo insertion of a nasogastric pH probe for assessment of gastric pH during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, 2-period, fixed-sequence study.
Groups:
- Baricitinib + Omeprazole: 10 milligram (mg) baricitinib tablet administered orally, once, on Day 1 in Period 1 and on Day 10 in Period 2.
  40 mg omeprazole capsule administered orally, once daily (QD), for 8 days (Days 3 through 10) in Period 2.
Period: Period 1 (Day 1 Through Predose Day 3)
Arm/Group | Baricitinib + Omeprazole
Started | 30
Received Baricitinib | 30
Completed | 30
Not Completed | 0
Period: Period 2 (At Dosing Day 3 Through Day12)
Arm/Group | Baricitinib + Omeprazole
Started | 30
Received Baricitinib | 30
Received 8 Doses of Omeprazole | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib + Omeprazole: 10 mg baricitinib tablet administered orally, once, on Day 1 in Period 1 and on Day 10 in Period 2.
  40 mg omeprazole capsule administered orally, QD, for 8 days (Days 3 through 10) in Period 2.
Arm/Group | Baricitinib + Omeprazole
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Baricitinib
Time Frame: Days 1 and 10: predose of baricitinib, 0.5, 0.75, 1, 2, 3, 4, 6, 12, 24, 36 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + omeprazole in Period 2) and had PK data to calculate Cmax of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Baricitinib: 10 mg baricitinib tablet administered orally, once, on Day 1 in Period 1.
- Baricitinib + Omeprazole: 10 mg baricitinib tablet administered orally, once, on Day 10 in Period 2.
  40 mg omeprazole capsule administered orally, QD, for 8 days (Days 3 through 10) in Period 2.
Arm/Group | Baricitinib | Baricitinib + Omeprazole
Number analyzed (Participants) | 30 | 30
nanograms/milliliter (ng/mL) | 99.2 (32) | 76.8 (25)

2. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Baricitinib
Time Frame: Days 1 and 10: predose of baricitinib, 0.5, 0.75, 1, 2, 3, 4, 6, 12, 24, 36 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + omeprazole in Period 2) and had PK data to calculate Tmax of baricitinib.
Measure: Median (Full Range); unit: hours
Arm/Group | Baricitinib | Baricitinib + Omeprazole
Number analyzed (Participants) | 30 | 30
hours | 1.00 [0.50 to 3.00] | 2.00 [0.75 to 6.00]

3. Primary Outcome: PK: Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity [AUC(0-∞)] of Baricitinib
Time Frame: Days 1 and 10: predose of baricitinib, 0.5, 0.75, 1, 2, 3, 4, 6, 12, 24, 36 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + omeprazole in Period 2) and had PK data to calculate AUC(0-∞) of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Baricitinib | Baricitinib + Omeprazole
Number analyzed (Participants) | 30 | 30
nanograms*hour/milliliter (ng*h/mL) | 663 (23) | 712 (23)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 24).
Groups:
- Baricitinib: 10 mg baricitinib tablet administered orally once, on Day 1 in Period 1.
  Adverse events are reported from baseline through predose on Day 3.
- Omeprazole: 40 mg omeprazole capsule administered orally, QD, on Days 3 through 9 in Period 2.
  Adverse events are reported from postdose on Day 3 through predose on Day 10.
- Baricitinib + Omeprazole: 10 mg baricitinib tablet administered orally once with 40 mg omeprazole capsule orally once, on Day 10 in Period 2.
  Adverse events are reported from postdose on Day 10 up to Day 24.
Arm/Group | Baricitinib | Omeprazole | Baricitinib + Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 8/30 | 7/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=30) | Omeprazole (N=30) | Baricitinib + Omeprazole (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days